CLINICAL TRIAL: NCT03431181
Title: Optimal VAsopressor TitraTION in Patients 65 Years and Older (OVATION-65)
Brief Title: Optimal VAsopressor TitraTION in Patients 65 Years and Older
Acronym: OVATION-65
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, François Lamontagne, Doctor, professor and researcher, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MP-31-2018-1789
Record Dates: First submitted 2018-02-04; First posted 2018-02-13 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Vasopressors; Hypotension; Mean Arterial Pressure Targets; Usual Care
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAP target 60-65 mmHg (Experimental): Treating teams will adjust vasopressors to a target MAP range of 60 to 65 mmHg, avoiding vasopressor-induced MAP above this range.
  Interventions: Behavioral: MAP target 60-65 mmHg
- Usual Care (Active Comparator): Patients in the control arm will receive usual care (as per local practices).
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: MAP target 60-65 mmHg — Treating teams will adjust vasopressors to a target MAP range of 60 to 65 mmHg, avoiding vasopressor-induced MAP above this range.
  Arms: MAP target 60-65 mmHg
Behavioral: Usual care — Patients in the control arm will receive usual care (as per local practices).
  Arms: Usual Care

SUMMARY:
We have designed OVATION-65 to evaluate the effects of permissive low blood pressure compared to usual care on markers of organ injury and survival in older patients.

DETAILED DESCRIPTION:
Background:

When it is severe, hypotension compromises tissue perfusion and organ function, leading to multiple organ failure and death. Commonly in intensive care units (ICUs), excessive vasodilation causes hypotension. In response, clinicians administer vasopressors to induce vasoconstriction and thereby raise blood pressure. However, these medications may reduce blood flow to vital organs, including the heart, and therefore damage them. Titrating vasopressors therefore requires balancing the risks of organ dysfunction arising from vasopressors or hypotension. Current guidelines recommend titrating vasopressors to a mean arterial pressure (MAP) of 65 mmHg. By not specifying an upper limit, guidelines and clinicians put more emphasis on preventing hypotension than on minimizing vasopressor exposure. Permissive hypotension, defined as a MAP target below traditional levels, may reduce vasopressor-induced harm while avoiding organ dysfunction induced by severe hypotension.

Observational data show that the average MAP in Canadian patients on vasopressors is 75 mmHg, 10 mmHg above current guideline recommendations and self-reported practices.The recent CIHR-funded OVATION pilot RCT (n=118) of permissive hypotension met feasibility objectives of demonstrating a separation in mean MAP between arms (9 mmHg, p<0.0001) and enrolling patients efficiently (2.3 patients/site/month). Investigators have also completed an individual patient data meta-analysis with the French SEPSISPAM trial and found that a lower MAP target may be beneficial in patients 65 years old.

Objective:

The overarching goal of this randomized controlled trial (RCT) of permissive hypotension vs. usual blood pressure targets in hypotensive patients ≥65 years old is to determine whether permissive hypotension reduces the risk of harm associated with usual vasopressor therapy. The proposed RCT has specific objectives to ascertain the effect of permissive hypotension vs. usual care on: 1) markers of organ injury (primarily in the heart at day 3, secondarily (on day 3 and day 7) in the brain, liver, intestine, and skeletal muscle); 2) global tissue dysoxia (assessed by plasma lactate); 3) organ function (assessed by Sequential Organ Failure Assessment [SOFA] Score ); 4) resource utilization, 5) pre-specified adverse events, 6) mortality at 90 days and 6 months; 7) cognitive impairment in survivors at 6 months.

Methods:

Eligible patients will be randomized to target MAP 60-65 mmHg vs. usual care. By comparing permissive hypotension to usual care, we improve acceptance from clinicians and reduce the risk that the control group will diverge widely from usual care. Investigators will enroll patients in 7 Canadian ICUs. The deferred consent model will be adopted, successfully used in the pilot trial. Risk of bias will be minimized by allocation concealment, blinding of outcome assessors, complete hospital follow-up and intention-to-treat analysis.

Relevance:

This RCT proposal is embedded in the international OVATION-65 program of research, which includes the ongoing NIHR-funded UK65 Trial which measures 90-day mortality as the primary outcome. The Canadian OVATION-65 RCT is the only trial that measures organ injury biomarkers, providing crucial clinical information regardless of the effect on mortality. Results are expected to be incorporated into guidelines to inform practice worldwide.

Sample size:

The OVATION-65 Trial was designed to be complementary to the 65 Trial conducted in the United Kingdom. The original proposal, which consisted in a larger and simpler trial (n=800 participants, focused on biomarkers of organ injury) was abandoned because funding applications to the Canadian Institutes for Health Research and the Canadian Frailty Network were unsuccessful. The current trial was supported by a combination of multiple more modest operating grants awarded by the Université de Sherbrooke and the Centre de Recherche du CHU de Sherbrooke (see Funding sources). However, each grant required a distinct objective increasing the complexity of the analysis plan and sample size calculation. Certain analyses were incorporated into funding applications for local experiments on a small scale. By combining funds from multiple sources, we are able to enroll up to 200 participants, however we lack resources to measure every outcome on 200 participants. Outcomes that cannot be measured on every participant or as well as those that were planned originally but that remain unfunded are described briefly in the secondary outcomes section and specified as ancillary studies. They will be reported separately.

Attempts to obtain funding for a larger OVATION-65 Trial continued until the end of 2018. Sufficient funding was secured to enroll up to 200 patients, but trial enrollment was terminated on 21 February 2020 after 159 patients were enrolled, on the recommendation of the DSMC following publication of the 65 trial. Six-month follow-up will be complete in August 2020. The statistical analysis plan will be registered and published before analyzing the data.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or older
2. Working diagnosis of vasodilatory hypotension as assessed by treating team
3. Vasopressors started for 12 hours or less (window from ICU admission after/during adequate fluid resuscitation as assessed by treating physician)
4. Vasopressors expected for 6 additional hours as assessed by the treating team

Exclusion Criteria:

1. Actively treated for spinal cord injury or acute brain injury
2. Vasopressors being given solely for bleeding, acute ventricular failure or post-cardiopulmonary bypass vasoplegia
3. Lacking commitment to life-sustaining therapies (expected withdrawal of life-sustaining treatments within the next 48 hours
4. Death perceived as imminent
5. Previously enrolled in OVATION-65
6. Organ transplant within the last year
7. Extra corporeal life support at baseline
8. The treating physician(s) lacks equipoise regarding the overall effects of permissive hypotension versus usual care on patient important outcomes.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 159 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma high-sensitivity cardiac troponin T at day 3 (primary mechanistic outcome) | Day 3
  Plasma high-sensitivity cardiac troponin T (hsTnT) at day 3 (corrected for baseline levels) (primary mechanistic outcome)

SECONDARY OUTCOMES:
Concentration of biomarkers associated with tissue injury to the brain | Days 1 (baseline),3 and 7
  Concentration of biomarkers associated with tissue injury to the brain (plasma GFAP, plasma Myelin Basic Protein and serum NSE)
Concentration of biomarker associated with tissue injury to the liver | Days 1 (baseline),3 and 7
  Concentration of biomarker associated with tissue injury to the liver (plasma ALT)
Concentration of biomarker associated with tissue injury to the intestine | Days 1 (baseline),3 and 7
  Concentration of biomarker associated with tissue injury to the intestine (plasma fatty acid binding protein (FABP))
Concentration of biomarker associated with tissue injury to the skeletal muscle | Days 1 (baseline),3 and 7
  Concentration of biomarker associated with tissue injury to the skeletal muscle (plasma creatinine kinase).
Concentration of biomarker associated with cardiac wall stress | Days 1 (baseline),3 and 7
  Concentration of biomarker associated with cardiac wall stress (plasma N-terminal pro-B-type natriuretic peptide [NT-proBNP]).
Global tissue dysoxia | Days 1 (baseline),3 and 7
  Global tissue dysoxia will be assessed through plasma lactate
Plasma high-sensitivity cardiac troponin T (hsTnT) | Day 7
  Plasma high-sensitivity cardiac troponin T (hsTnT) at day 7
Pre-specified adverse events | 28 days
  Pre-specified adverse events assessed by events of stroke, clinically detected supraventricular arrhythmia, acute kidney injury (KDIGO stage 3), limb or intestinal ischemia
Organ function | Days 1 (baseline), 2, 3, 4, 7, 10, 14 and 28
  Organ function using SOFA score (measured at baseline (day 1) and on days 2,3,4,7,10,14 and 28 while in the ICU)
Mortality | 90 days and 6 months
  Mortality at 90 days and at 6 months will be assessed during the phone call at 6 months
6-month cognitive impairment | 6 months
  6-month cognitive impairment assessed by Telephone Interview for Cognitive Status (TICS)
Healthcare utilization | 28 days
  Healthcare utilization assessed by measuring duration of mechanical ventilation, renal replacement therapy, vasopressor therapy and ICU and hospital stay (through days of utilization)
Plasma level of ascorbic acid (outcome for ancillary study) | Day 1 (baseline)
  Plasma level of ascorbic acid (measured at baseline (day 1))
Biomarkers of ascorbic acid deficiency-related organ injury (outcome for ancillary study) | Days 1 (baseline), 3 and 7
  Inflammation (IL-1ß; TNF-α; CRP) and endothelial injury (thrombomodulin, angiopoietin-2)
Discovery proteomic approach to identify peptides and proteins expressed in the urine (outcome for ancillary study) | Days 1 (baseline), 3 and 7
  Discovery proteomic approach through novel urine biomarkers
Validate the predictive value of five prespecified biomarkers of renal injury in urine using a proteomic approach (outcome for ancillary study): TIMP2, NGAL, FABPL, CYTC, IGFBP7 | Days 1 (baseline), 3 and 7
  Proteomic discovery approach through validation of prespecified urine biomarkers: TIMP2, NGAL, FABPL, CYTC, IGFBP7
Impact of vasopressor regimen on the immune response, adrenergic receptor activity and related proteomic signature of peripheral blood mononuclear cell (PBMC) (outcome for ancillary study) | Day 1 (baseline) and 7
  Immune response, adrenergic receptor activity and proteomic profile through Th1/Th2 profiling, PBMC adrenergic receptors AMPc activity and proteomic signature and associations with responses to catecholamines.

CONTACTS AND LOCATIONS:
Overall Officials: François Lamontagne, MD FRCPC MSc, Principal Investigator — University of Sherbrooke and CIUSSS de l'Estrie-CHUS; Neill Adhikari, MDCM MSc, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto
Locations (1):
- CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Masse MH, Battista MC, Wilcox ME, Pinto R, Marinoff N, D'Aragon F, St-Arnaud C, Mayette M, Leclair MA, Quiroz Martinez H, Grondin-Beaudoin B, Poulin Y, Carbonneau E, Seely AJE, Watpool I, Porteous R, Chasse M, Lebrasseur M, Lauzier F, Turgeon AF, Bellemare D, Mehta S, Charbonney E, Belley-Cote E, Botton E, Cohen D, Lamontagne F, Adhikari NKJ; OVATION-65 team members; Canadian Critical Care Trials Group. Optimal VAsopressor TitraTION in patients 65 years and older (OVATION-65): protocol and statistical analysis plan for a randomised clinical trial. BMJ Open. 2020 Nov 14;10(11):e037947. doi: 10.1136/bmjopen-2020-037947. PMID 33191251